CLINICAL TRIAL: NCT03691662
Title: A Phase III, Randomized, Double-Masked, Active-Controlled, Parallel-Group, Multicenter Study Assessing the Efficacy and Safety of DE-117 Ophthalmic Solution Compared With Timolol Maleate Ophthalmic Solution 0.5% in Subjects With Glaucoma or Ocular Hypertension - Spectrum 4 Study
Brief Title: A Phase III Study Assessing the Efficacy and Safety of DE-117 Ophthalmic Solution Compared With Timolol Maleate Ophthalmic Solution 0.5% in Subjects With Glaucoma or Ocular Hypertension - Spectrum 4 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 011710IN
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Results first posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Glaucoma and Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DE-117 Ophthalmic Solution (Experimental): Topical DE-117 Ophthalmic Solution once daily and Vehicle once daily for 3 months
  Interventions: Drug: DE-117 Ophthalmic Solution
- Timolol Maleate Ophthalmic Solution 0.5% (Active Comparator): Topical Timolol Maleate Ophthalmic Solution 0.5% twice daily for 3 months
  Interventions: Drug: Timolol Maleate Ophthalmic Solution 0.5%

INTERVENTIONS:
Drug: DE-117 Ophthalmic Solution — Topical DE-117 Ophthalmic Solution once daily and Vehicle once daily for 3 months
  Arms: DE-117 Ophthalmic Solution
Drug: Timolol Maleate Ophthalmic Solution 0.5% — Topical Timolol Maleate Ophthalmic Solution 0.5% twice daily for 3 months
  Arms: Timolol Maleate Ophthalmic Solution 0.5%

SUMMARY:
This is a Phase III, randomized, double-masked, active-controlled, parallel-group, multi-center study. Subjects diagnosed with glaucoma or OHT who meet eligibility criteria at Visit 1 (Screening) will washout of their current topical IOP-lowering medication(s), if any. After completing the required washout period, subjects will return for Visit 2 (Baseline, Day 1). Subjects who meet all eligibility criteria at baseline will be randomized to receive double-masked treatment for 3 months.

Approximately 400 adult subjects and up to 30 pediatric subjects with glaucoma or OHT who meet all eligibility criteria will be randomized in a 1:1 ratio to receive either:

* DE-117 Ophthalmic Solution once daily and Vehicle once daily, or
* Timolol Maleate Ophthalmic Solution 0.5% twice daily. The study will evaluate the efficacy and safety of DE-117 Ophthalmic Solution compared with Timolol Maleate Ophthalmic Solution 0.5% in subjects with glaucoma or OHT through Month 3.

ELIGIBILITY:
Inclusion Criteria:

• glaucoma or ocular hypertension

Exclusion Criteria:

* Females who are pregnant, nursing, or planning a pregnancy
* Any corneal abnormality or other condition interfering with or preventing reliable tonometric measurements

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Arizona Eye Center, Chandler, Arizona
  - M & M Eye Institute, Prescott, Arizona
  - Global Research Management, Glendale, California
  - United Medical Research Inst, Inglewood, California
  - Eye Research Foundation, Newport Beach, California
  - North Bay Eye Associates Inc., Petaluma, California
  - Sacramento Eye Consultants, Sacramento, California
  - AdvanceMed Clinical Research, San Diego, California
  - Michael K. Tran, MD, Inc., Westminster, California
  - Haas Vision Center, Colorado Springs, Colorado
  - Florida Ophthalmic Institute, Gainesville, Florida
  - St. Michaels Eye Laser Institute, Largo, Florida
  - International Eye Associates PA, Ormond Beach, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Clayton Eye Clinical Research, LLC, Morrow, Georgia
  - Seidenberg Protzko Eye Associates, Havre de Grace, Maryland
  - Great Lakes Eye Care P.C, Saint Joseph, Michigan
  - Discover Vision Centers, Independence, Missouri
  - Silverstein Eye Centers, Kansas City, Missouri
  - Comprehensive Eye Care Ltd., Washington, Missouri
  - AdvanceMed Clinical Research, Las Vegas, Nevada
  - Rochester Ophthalmological Group, PC, Rochester, New York
  - Asheville Eye Associates, Asheville, North Carolina
  - Abrams Eye Center, Cleveland, Ohio
  - Total Eye Care PA, Memphis, Tennessee
  - VRF Eye Specialty Group, Memphis, Tennessee
  - Glaucoma Associates of Texas, Dallas, Texas
  - Houston Eye Associates HEA - Gramercy Location, Houston, Texas
  - Baylor College of Medicine Alkek Eye Center, Houston, Texas
  - The Eye Clinic of Texas, League City, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Stacy R. Smith M.D. P.C., Salt Lake City, Utah
  - Vistar Eye Center, Roanoke, Virginia
  - Tidewater Clinical Research, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DE-117 Ophthalmic Solution 0.002% QD (20:00) and Vehicle QD (08:00): DE-117 0.002% QD in the evening (20:00) and vehicle QD in the morning (08:00).
- Timolol Maleate Ophthalmic Solution 0.5% BID (20:00 & 08:00): Timolol Maleate Ophthalmic Solution 0.5% Twice a day (20:00 & 08:00)
Period: Overall Study
Arm/Group | DE-117 Ophthalmic Solution 0.002% QD (20:00) and Vehicle QD (08:00) | Timolol Maleate Ophthalmic Solution 0.5% BID (20:00 & 08:00)
Started | 208 | 209
Safety and Full Analysis Set (FAS) Participants | 204 (4 Participants did not receive DE-117 study drug.) | 205 (4 Participants did not receive Timolol.)
Completed | 187 | 196
Not Completed | 21 | 13

BASELINE CHARACTERISTICS:
Population: The Baseline Participants are similar in count to the Safety and Full Analysis Set (FAS) Participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | DE-117 Ophthalmic Solution 0.002% QD (20:00) and Vehicle QD (08:00) | Timolol Maleate Ophthalmic Solution 0.5% BID (20:00 & 08:00) | Total
Number analyzed (Participants) | 204 | 205 | 409
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 87 | 176
  >=65 years | 115 | 118 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (11.43) | 64.8 (11.56) | 64.4 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 109 | 230
  Male | 83 | 96 | 179
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 8 | 8 | 16
  Black or African American | 72 | 54 | 126
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 122 | 140 | 262
  Other | 0 | 0 | 0
  Multiple | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 204 | 205 | 409

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) at Week 1
Description: Intraocular Pressure: Analysis of IOP Score using Mixed Model for Repeated Measures (MMRM) on Observed Cases (Study Eye, Full Analysis Set). Intraocular Pressure (IOP), the fluid pressure inside the eye was measured with calibrated Goldmann applanation tonometer in millimeters mercury (mmHg) at 3 time points throughout the day.
Time Frame: 08:00, 10:00 and 16:00 at Week 1
Population: Full Analysis Set (FAS) included all randomized subjects who received at least one dose of study medication and provided baseline and at least one post-baseline IOP measurement. The number of analyzed are participants evaluable for the outcome measure at Week 1.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution 0.002% QD (20:00) and Vehicle QD (08:00) | Timolol Maleate Ophthalmic Solution 0.5% BID (20:00 & 08:00)
Number analyzed (Participants) | 204 | 205
mmHg
  8:00: number analyzed (Participants) | 202 | 203
  8:00 | 19.4 (0.23) | 19.7 (0.23)
  10:00: number analyzed (Participants) | 201 | 203
  10:00 | 18.5 (0.22) | 18.9 (0.22)
  16:00: number analyzed (Participants) | 198 | 200
  16:00 | 17.9 (0.23) | 18.6 (0.22)

2. Primary Outcome: Intraocular Pressure (IOP) at Week 6
Description: as for outcome 1
Time Frame: 08:00, 10:00 and 16:00 at Week 6
Population: Full Analysis Set (FAS) included all randomized subjects who received at least one dose of study medication and provided baseline and at least one post-baseline IOP measurement. The number of analyzed are participants evaluable for the outcome measure at Week 6.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution 0.002% QD (20:00) and Vehicle QD (08:00) | Timolol Maleate Ophthalmic Solution 0.5% BID (20:00 & 08:00)
Number analyzed (Participants) | 204 | 205
mmHg
  8:00: number analyzed (Participants) | 194 | 199
  8:00 | 20.4 (0.22) | 19.5 (0.21)
  10:00: number analyzed (Participants) | 194 | 198
  10:00 | 19.5 (0.20) | 18.8 (0.20)
  16:00: number analyzed (Participants) | 193 | 197
  16:00 | 19.2 (0.21) | 18.8 (0.21)

3. Primary Outcome: Intraocular Pressure (IOP) at Month 3
Description: as for outcome 1
Time Frame: 08:00, 10:00 and 16:00 at Month 3
Population: Full Analysis Set (FAS) included all randomized subjects who received at least one dose of study medication and provided baseline and at least one post-baseline IOP measurement. The number of analyzed are participants evaluable for the outcome measure at Month 3.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution 0.002% QD (20:00) and Vehicle QD (08:00) | Timolol Maleate Ophthalmic Solution 0.5% BID (20:00 & 08:00)
Number analyzed (Participants) | 204 | 205
mmHg
  8:00: number analyzed (Participants) | 189 | 197
  8:00 | 20.0 (0.22) | 19.6 (0.22)
  10:00: number analyzed (Participants) | 188 | 197
  10:00 | 19.4 (0.23) | 18.9 (0.22)
  16:00: number analyzed (Participants) | 188 | 197
  16:00 | 19.1 (0.23) | 19.0 (0.22)

4. Secondary Outcome: Mean Diurnal Intraocular Pressure (IOP) at Month 3 (First Key Secondary Endpoint)
Description: To determine if the mean diurnal IOP reduction with DE-117 ophthalmic solution 0.002% is superior to that of Timolol Maleate ophthalmic solution 0.5% at Month 3 in subjects with OAG or OHT. Mean Diurnal IOP is defined as the average IOP of all three timepoints (8AM, 10AM and 4PM) at Month 3.
Time Frame: Month 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution 0.002% QD (20:00) and Vehicle QD (08:00) | Timolol Maleate Ophthalmic Solution 0.5% BID (20:00 & 08:00)
Number analyzed (Participants) | 188 | 197
mmHg | 19.5 (0.19) | 19.2 (0.19)

5. Secondary Outcome: Intraocular Pressure (IOP) at Week 1 With Baseline Mean Diurnal IOP Less Than 25 mmHg (Second Key Secondary Endpoint)
Description: Intraocular Pressure (IOP) at Week 1 with baseline mean diurnal IOP less than 25 mmHg (Second Key Secondary Endpoint)
Time Frame: 08:00, 10:00 and 16:00 at week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution 0.002% QD (20:00) and Vehicle QD (08:00) | Timolol Maleate Ophthalmic Solution 0.5% BID (20:00 & 08:00)
Number analyzed (Participants) | 112 | 128
mmHg
  8:00 | 18.3 (0.28) | 19.1 (0.26)
  10:00: number analyzed (Participants) | 111 | 127
  10:00 | 17.5 (0.27) | 18.2 (0.25)
  16:00: number analyzed (Participants) | 109 | 126
  16:00 | 17.0 (0.27) | 18.0 (0.25)

6. Secondary Outcome: Intraocular Pressure (IOP) at Week 6 With Baseline Mean Diurnal IOP Less Than 25 mmHg (Second Key Secondary Endpoint)
Description: Intraocular Pressure (IOP) at Week 6 with baseline mean diurnal IOP less than 25 mmHg (Second Key Secondary Endpoint)
Time Frame: 08:00, 10:00 and 16:00 at week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution 0.002% QD (20:00) and Vehicle QD (08:00) | Timolol Maleate Ophthalmic Solution 0.5% BID (20:00 & 08:00)
Number analyzed (Participants) | 112 | 128
mmHg
  8:00: number analyzed (Participants) | 109 | 123
  8:00 | 19.4 (0.28) | 18.9 (0.26)
  10:00: number analyzed (Participants) | 109 | 122
  10:00 | 18.6 (0.25) | 18.2 (0.24)
  16:00: number analyzed (Participants) | 109 | 121
  16:00 | 18.4 (0.26) | 18.0 (0.24)

7. Secondary Outcome: Intraocular Pressure (IOP) at Month 3 With Baseline Mean Diurnal IOP Less Than 25 mmHg (Second Key Secondary Endpoint)
Description: Intraocular Pressure (IOP) at Month 3 with baseline mean diurnal IOP less than 25 mmHg (Second Key Secondary Endpoint)
Time Frame: 08:00, 10:00 and 16:00 at month 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution 0.002% QD (20:00) and Vehicle QD (08:00) | Timolol Maleate Ophthalmic Solution 0.5% BID (20:00 & 08:00)
Number analyzed (Participants) | 112 | 128
mmHg
  8:00: number analyzed (Participants) | 106 | 121
  8:00 | 18.9 (0.29) | 18.8 (0.27)
  10:00: number analyzed (Participants) | 106 | 121
  10:00 | 18.3 (0.28) | 18.0 (0.26)
  16:00: number analyzed (Participants) | 106 | 121
  16:00 | 18.1 (0.28) | 18.0 (0.26)

8. Secondary Outcome: Mean Diurnal Intraocular Pressure (IOP) at Week 1 (Third Key Secondary Endpoint)
Description: The third key secondary endpoint, mean diurnal IOP at Week 1, the hypothesis of superiority of DE-117 to timolol was tested. Analysis using MMRM on Observed Cases.
  Mean Diurnal IOP is defined as the average IOP of all three timepoints (8AM, 10AM and 4PM) at week 1.
Time Frame: week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-117 Ophthalmic Solution 0.002% QD (20:00) and Vehicle QD (08:00) | Timolol Maleate Ophthalmic Solution 0.5% BID (20:00 & 08:00)
Number analyzed (Participants) | 198 | 200
mmHg | 18.6 (0.20) | 19.1 (0.20)

ADVERSE EVENTS:
Time Frame: Adverse events in this study were collected from the time of informed consent and were followed to resolution, or until the subject's participation in the study ended at Month 3.
Description: The safety population includes all randomized participants who received at least one dose of the study medication and similar in count to the Full Analysis Set population.
  Other Adverse events data is a summary of AEs observed at a rate of 1.0% or higher by System Organ Class and Preferred Term. Threshold of 0.98% is considered 1% and therefore added.
Arm/Group | DE-117 Ophthalmic Solution | Timolol Maleate Ophthalmic Solution 0.5%
All-Cause Mortality (participants affected / at risk) | 1/204 | 0/205
Serious Adverse Events (participants affected / at risk) | 7/204 | 1/205
Other Adverse Events (participants affected / at risk) | 68/204 | 49/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DE-117 Ophthalmic Solution (N=204) | Timolol Maleate Ophthalmic Solution 0.5% (N=205)
Cystoid macular oedema (Eye disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DE-117 Ophthalmic Solution (N=204) | Timolol Maleate Ophthalmic Solution 0.5% (N=205)
Conjunctival hyperaemia (Eye disorders) | 16 | 7
Photophobia (Eye disorders) | 12 | 1
Vision blurred (Eye disorders) | 6 | 2
Ocular hyperaemia (Eye disorders) | 4 | 2
Anterior chamber cell (Eye disorders) | 3 | 0
Cystoid macular oedema (Eye disorders) | 2 | 0
Erythema of eyelid (Eye disorders) | 2 | 2
Eye pain (Eye disorders) | 4 | 2
Growth of eyelashes (Eye disorders) | 2 | 5
Iritis (Eye disorders) | 2 | 0
Ocular discomfort (Eye disorders) | 2 | 0
Dry eye (Eye disorders) | 2 | 2
Eye pruritus (Eye disorders) | 2 | 0
Lacrimation increased (Eye disorders) | 2 | 0
Punctate keratitis (Eye disorders) | 2 | 1
Visual impairment (Eye disorders) | 2 | 3
Instillation site pain (General disorders) | 11 | 13
Intraocular pressure increased (Investigations) | 5 | 0
Vital dye staining cornea present (Investigations) | 2 | 1
Vitreous detachment (Eye disorders) | 3 | 1
Conjunctival haemorrhage (Eye disorders) | 2 | 3
Foreign body sensation in eyes (Eye disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 3
Bronchitis (Infections and infestations) | 2 | 3
Influenza (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 0 | 3
Blood pressure increased (Investigations) | 2 | 0
Headache (Nervous system disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT03691662/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT03691662/SAP_001.pdf